CLINICAL TRIAL: NCT00051129
Title: An Evaluation of Safety and Efficacy of Anecortave Acetate Versus Placebo in Patients With Subfoveal Choroidal Neovascularization Due to Exudative Age-Related Macular Degeneration.
Brief Title: Anecortave Acetate in Subfoveal Choroidal Neovascularization (CNV) Due to Wet Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-27
Record Dates: First submitted 2003-01-03; First posted 2003-01-07 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2008-08

CONDITIONS: Macular Degeneration; Maculopathy, Age-Related; Age-Related Maculopathies; Age-Related Maculopathy; Maculopathies, Age-Related
Keywords: AMD; anecortave acetate; wet AMD; age-related macular degeneration; Macular Degeneration; Maculopathy, Age-Related; Age-Related Maculopathies; Age-Related Maculopathy; Maculopathies, Age-Related
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Anecortave Acetate (Experimental): Posterior juxtascleral injection in the study eye at 6 month intervals (Day 0, Month 6, Month 12, Month 18)
  Interventions: Drug: Anecortave Acetate 15 mg sterile suspension
- Anecortave Acetate Vehicle (Placebo Comparator): Posterior juxtascleral injection in the study eye at 6 month intervals (Day 0, Month 6, Month 12, Month 18)
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate 15 mg sterile suspension — 0.5 ml of 30 mg/ml administered as a posterior juxtascleral injection
  Arms: Anecortave Acetate
Other: Anecortave Acetate Vehicle — Administered as a posterior juxtascleral injection
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study was to evaluate anecortave acetate compared to placebo for maintenance of visual acuity after 24 months of treatment in patients with subfovial choroidal neovascularization (CNV) due to exudative age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of exudative AMD and a primary or recurrent subfoveal CNV lesion in the study eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 50 years.
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in logMAR visual acuity score at 12 months | Month 12